CLINICAL TRIAL: NCT00461058
Title: A Randomized, Double Blind Study to Compare the Safety and Tolerability of Aleglitazar and Actos in Patients With Type 2 Diabetes and NYHA Class II Heart Failure.
Brief Title: A Comparative Study of Aleglitazar and Actos in Patients With Type 2 Diabetes Mellitus and New York Heart Association (NYHA) Class II Heart Failure.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC20265
Record Dates: First submitted 2007-04-16; First posted 2007-04-17 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; aleglitazar

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Actos (Active Comparator)
  Interventions: Drug: Actos
- Aleglitazar (Experimental)
  Interventions: Drug: aleglitazar

INTERVENTIONS:
Drug: Actos — Titrated to an individual maximum tolerated dose up to 45mg p.o. daily
  Arms: Actos
Drug: aleglitazar — Titrated to an individual maximum tolerated dose up to 0.3mg p.o. daily
  Arms: Aleglitazar

SUMMARY:
This 2 arm study will compare the safety, tolerability and efficacy of aleglitazar and Actos in patients with type 2 diabetes and symptomatic NYHA class II heart failure. Eligible patients will be randomized to receive either aleglitazar, titrated to an individual maximum tolerated dose up to 0.3mg p.o. daily, or Actos, titrated to an individual maximum tolerated dose up to 45mg p.o. daily, in addition to prescribed diabetes therapy where applicable. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* type 2 diabetes for >=1 month;
* drug naive, or receiving stable doses of <=2 oral antihyperglycemic medications;
* HbA1c 6.5-10.0% at screening;
* symptomatic, stable NYHA class 2 heart failure at screening.

Exclusion Criteria:

* type 1 diabetes;
* current or previous treatment with insulin;
* uncontrolled hypertension;
* NYHA class 1, 3 or 4 at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Incidence of cardiovascular death, hospitalization or clinic visit for heart failure with i.v. administration of diuretics during 26 week treatment period. | 26 week

SECONDARY OUTCOMES:
Safety: peripheral oedema, deterioration of heart failure, increase in body weight during 26 week treatment period, adverse events (AEs), laboratory parameters. | 26 week
Efficacy: Change from baseline to week 26 in Hemoglobin A1c (HbA1c), fasting plasma glucose (FPG), fasting plasma insulin (FPI) and lipid profile. | 26 week

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- United States (10):
  - Jonesboro, Arkansas
  - Carmichael, California
  - Loma Linda, California
  - Long Beach, California
  - Jacksonville, Florida
  - Slidell, Louisiana
  - Minneapolis, Minnesota
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
- Israel (3):
  - Ashkelon
  - Haifa
  - Kfar Saba
- Mexico (7):
  - Culiacán
  - Guadalajara
  - Metepec
  - Mexico City
  - Monterrey
  - Pachuca
  - San Luis Potosí City
- Romania (7):
  - Arad
  - Bacau
  - Baia Mare
  - Bucharest
  - Oradea
  - Ploieşti
  - Târgovişte
- Russia (4):
  - Moscow
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Ukraine (3):
  - Donetsk
  - Kharkiv
  - Kiev